CLINICAL TRIAL: NCT02110381
Title: Assessing Alternative Approaches for Blood Pressure Control: A3BC Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was a pilot study and we enrolled sufficient numbers to evaluate the proposed outcomes.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elizabeth A. Jackson, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00086973
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: High blood pressure
MeSH Terms: conditions — Hypertension

ARMS (2):
- Device Guided Breathing/Combination Therapy (Active Comparator): Participants will first do device guided breathing for 8 weeks, followed by 8 weeks of doing BOTH the device guided breathing AND the hand grip exercises. Participants will be given a home blood pressure monitor. Participants will measure blood pressure and heart rate at home for 2 weeks prior to starting any intervention and also during the 16 week of intervention.
  Interventions: Device: Device guided breathing RESPeRATE; Device: Isometric hand grip Zona Plus
- Isometric Hand Grip/Combination Therapy (Active Comparator): Participants will first do isometric hand grip exercises for 8 weeks, followed by 8 weeks of doing BOTH the device guided breathing AND the hand grip exercises. Participants will be given a home blood pressure monitor. Participants will measure blood pressure and heart rate at home for 2 weeks prior to starting any intervention and also during the 16 week of intervention.
  Interventions: Device: Device guided breathing RESPeRATE; Device: Isometric hand grip Zona Plus

INTERVENTIONS:
Device: Device guided breathing RESPeRATE — Participants will use a device called RESPeRATE which will measure how many breaths they take per minute. A strap wraps around the participants chest that measures breathing frequency. Headphones plug into the device to inform participants about their breathing. The device will help guide participants to breathe slowly using musical tones, with a goal of about ten breaths per minute.
  Participants will use the breathing device 5 days per week for about 15 minutes each day. Participants will keep a log of their exercises and return it with each visit.
Device: Isometric hand grip Zona Plus — Participants will use a device called the Zona Plus, which they will hold in their hand and squeeze. A session consists of 2 minutes of squeezing the device followed by 1 minute of rest. Participants will do a total of 4 sessions (2 sessions for each hand) for a total of about 12 minutes of exercise.
  Participants will do these exercises 5 days per week. Participants will keep a log of their exercise and return it with each visit.

SUMMARY:
An estimated 76 million adults in the United States over the age of 20 have hypertension (HTN); which translates into 1 out of 3 adults. Globally the prevalence of HTN is over 25% for adults, and accounts for approximately 13.5% of all deaths. Given the aging of the population together with increases in obesity and sedentary behavior, it is not surprising that HTN is projected to increase significantly over the next several decades; with over 1.5 billion adults having HTN by the year 2025. Thus the public health implications to preventing and/or reducing elevations in blood pressure are substantial.

This study compares the efficacy of two different non-pharmacologic interventions (device guided breathing and isometric hand grip exercises) used alone and in combination for lowering blood pressure. This pilot study will include 30 adults with stage 1 hypertension. The primary outcome is the change in blood pressure from baseline to 8 weeks. Secondary outcomes include change in blood pressure from 8 weeks to 16 weeks and acceptability of the interventions by participants. The knowledge gained from this study can provide information on non-pharmacologic methods that may be useful in decreasing blood pressure. Such knowledge may be especially useful for patients for whom access to medications and health care is limited and among patients unwilling to take or intolerant to pharmacologic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 21 years old, and
* Have Stage 1 high blood pressure. (Defined as a systolic blood pressure between 140 mm Hg and 159 mm Hg (the top blood pressure number) and/or a diastolic blood pressure between 90 mm Hg and 99 mm Hg (the bottom blood pressure number) in the prior 6 months.)

Exclusion Criteria:

* Take drugs to control blood pressure.
* Have a history of left ventricular hypertrophy.
* Have a history of cardiovascular disease such as stroke, mini-strokes, heart attack, unstable angina, bypass surgery, stents, angioplasty, abnormal heart rhythms, heart failure, or peripheral artery disease.
* Have diabetes.
* Have a history of poor kidney function.
* Have an upper arm circumference greater than 17 inches.
* Are currently participating in a formal exercise or weight loss program.
* Plan to participate in a formal exercise or weight loss program in the next 6 months.
* Are pregnant or plan to become pregnant in the next 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Jackson, MD MPH FACC, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical records were screened for initial eligibility criteria between 9/2014 - 4/2015. Patients were then contacted via letter and phone to gauge interest.
Pre-assignment Details: After consent, participants completed a run-in period in which they measured their blood pressure at home for 2 weeks. Participants with multiple readings greater than 160mmHg SBP or 100mmHg DBP were considered screen failures (n=13, plus 1 withdrawal).
Groups:
- Device Guided Breathing: Participants will first do device guided breathing for 8 weeks, followed by 8 weeks of doing BOTH the device guided breathing AND the hand grip exercises.
  Device guided breathing: Participants will use a device (RESPeRATE) to guide them through slow controlled breathing, with a goal of about ten breaths per minute.
  Participants will use the breathing device 5 days per week for about 15 minutes each day. Participants will keep a log of their exercises and return it with each visit.
  Isometric hand grip: Participants will use a device (Zona Plus) which they will hold in their hand and squeeze. A session consists of 2 minutes of squeezing followed by 1 minute of rest. Participants will do a total of 4 sessions (2 sessions for each hand) for a total of about 12 minutes of exercise.
  Participants will do these exercises 5 days per week. Participants will keep a log of their exercise and return it with each visit.
- Isometric Hand Grip: Participants will first do isometric hand grip exercises for 8 weeks, followed by 8 weeks of doing BOTH the hand grip exercises AND the device guided breathing.
  Isometric hand grip: Participants will use a device (Zona Plus) which they will hold in their hand and squeeze. A session consists of 2 minutes of squeezing followed by 1 minute of rest. Participants will do a total of 4 sessions (2 sessions for each hand) for a total of about 12 minutes of exercise.
  Participants will do these exercises 5 days per week. Participants will keep a log of their exercise and return it with each visit.
  Device guided breathing: Participants will use a device (RESPeRATE) to guide them through slow controlled breathing, with a goal of about ten breaths per minute.
  Participants will use the breathing device 5 days per week for about 15 minutes each day. Participants will keep a log of their exercises and return it with each visit.
Period: Single Modality
Arm/Group | Device Guided Breathing | Isometric Hand Grip
Started | 9 | 9
Completed | 7 | 8
Not Completed | 2 | 1
Period: Dual Modality
Arm/Group | Device Guided Breathing | Isometric Hand Grip
Started | 7 | 8
Began Active Treatment | 7 | 7
Completed | 5 | 7
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Guided Breathing | Isometric Hand Grip | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.75 (14.85) | 52.67 (15.48) | 54.59 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Systolic Blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 127.33 (10.15) | 133.57 (17.89) | 129.06 (9.00)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure
Description: Blood pressure was measured using an automated cuff with subject in a seated position for at least 5 minutes. Six measurements were recorded at 1-minute intervals. The mean was used in analysis.
Time Frame: 8 weeks and 16 weeks
Population: 9 subjects in each group were analyzed. These subjects represent the individuals who passed started the intervention phase of the study.
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Device Guided Breathing | Isometric Hand Grip
Number analyzed (Participants) | 9 | 9
mmHg (millimeters of mercury)
  Baseline Systolic Blood Pressure | 127.33 (10.15) | 133.57 (17.89)
  Change from baseline at 8-weeks | 5.71 (13.92) | 3.43 (8.00)
  Change from baseline at 16-weeks: number analyzed (Participants) | 4 | 6
  Change from baseline at 16-weeks | 3.50 (10.344) | 6.17 (12.30)

2. Secondary Outcome: Adherence to Single Modality Exercise (Device Guided Breathing or Isometric Hand Grip)
Description: Subjects recorded sessions on a log; they were expected to complete 5 days/week for 8 weeks of single modality exercise for a minimum of 40 reported sessions. Results are reported as number of subjects reporting a minimum of 40 sessions.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Device Guided Breathing | Isometric Hand Grip
Number analyzed (Participants) | 7 | 7
Participants | 7 | 4

3. Secondary Outcome: Adherence to Dual Modality Exercise (Device Guided Breathing + Isometric Hand Grip)
Description: as for outcome 2
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Device Guided Breathing | Isometric Hand Grip
Number analyzed (Participants) | 5 | 7
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: We were in contact with subjects for 18 weeks total.
Groups:
- Screen Failures: These subjects reflect individuals who: 1) consented to be in the study, 2) participated in the initial run-in period to evaluate blood pressure, 3) ended up not meeting the blood pressure criteria required for randomization
Arm/Group | Device Guided Breathing | Isometric Hand Grip | Screen Failures
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/9 | 1/9 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Guided Breathing (N=9) | Isometric Hand Grip (N=9) | Screen Failures (N=14)
High blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Blood pressure readings of greater than 200mmHg systolic blood pressure and/or greater than 100mmHg diastolic pressure
Tight blood pressure cuff (Investigations) | 0 (0) | 0 (0) | 1 (1) — Blood pressure cuff was too tight for subject comfort
Sore hands (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Musculoskeletal soreness from using the isometric handgrip device

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes